CLINICAL TRIAL: NCT06563999
Title: Neoadjuvant Umbrella Trial Directed by Next Generation Sequencing for Patients With Unresectable Stage III NSCLC Harboring Rare Mutations (Without EGFR Sensitizing Mutations)
Brief Title: Neoadjuvant Umbrella Trial for Patients With Unresectable Stage III NSCLC Harboring Rare Mutations.
Acronym: NUMER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Si-Yu Wang, Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-10117
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer Stage III; Mutation
Keywords: stage III NSCLC; rare mutations; umbrella trial; neoadjuvant
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Crizotinib; pralsetinib; larotrectinib; 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine; pyrotinib; ensartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Treatment 1-Sunvozertinib (Experimental): Patients with EGFR exon20ins mutation receive Sunvozertinib 300 mg orally once a day, 28 days as one cycle for 3 cycle.
  Interventions: Drug: Sunvozertinib
- Treatment 2-Crizotinib (Experimental): Patients with ROS1 fusion mutation receive Crizotinib 250mg orally once a day, 28 days as one cycle for 3 cycle.
  Interventions: Drug: Crizotinib
- Treatment 3-Pralsetinib (Experimental): Patients with RET fusion mutation receive Pralsetinib 400mg orally once a day, 28 days as one cycle for 3 cycle.
  Interventions: Drug: Pralsetinib
- Treatment 4-Larotrectinib (Experimental): Patients with NTRK fusion mutation receive Larotrectinib 100 mg orally twice daily, 28 days as one cycle for 3 cycle.
  Interventions: Drug: Larotrectinib
- Treatment 5-Savolitinib (Experimental): Patients with MET 14 exon mutation receive Savolitinib 600 mg or 400 mg (weight <50 kg) orally once a day, 28 days as one cycle for 3 cycle.
  Interventions: Drug: Savolitinib
- Treatment 6-Pyrotinib (Experimental): Patients with HER2 mutation receive Pyrotinib 400 mg orally once a day, 28 days as one cycle for 3 cycle.
  Interventions: Drug: Pyrotinib
- Treatment 7-Dabrafenib+Trametinib (Experimental): Patients with BRAF V600E mutation receive Dabrafenib plus Trametinib, 28 days as one cycle for 3 cycle.
  Interventions: Drug: Dabrafenib+Trametinib
- Treatment 8-Glecirasib (Experimental): Patients with KRAS G12C mutation receive Glecirasib 800 mg daily orally, 28 days as one cycle for 3 cycle.
  Interventions: Drug: Glecirasib
- Treatment 9-Ensartinib (Experimental): Patients with ALK fusion mutation receive Ensartinib 225 mg daily orally, 28 days as one cycle for 3 cycle.
  Interventions: Drug: Ensartinib

INTERVENTIONS:
Drug: Sunvozertinib — 300 mg orally once a day, 28 days as one cycle.
  Other Names: DZD9008
  Arms: Treatment 1-Sunvozertinib
Drug: Crizotinib — 300 mg orally once a day, 28 days as one cycle.
  Other Names: Xalkori
  Arms: Treatment 2-Crizotinib
Drug: Pralsetinib — 400 mg orally once a day, 28 days as one cycle.
  Other Names: GAVRETO
  Arms: Treatment 3-Pralsetinib
Drug: Larotrectinib — 100 mg orally twice daily, 28 days as one cycle.
  Other Names: VITRAKVI
  Arms: Treatment 4-Larotrectinib
Drug: Savolitinib — 600 mg or 400 mg (weight <50 kg) orally once a day, 28 days as one cycle.
  Other Names: ORPATHYS
  Arms: Treatment 5-Savolitinib
Drug: Pyrotinib — 400 mg orally once a day, 28 days as one cycle.
  Other Names: SHR1258
  Arms: Treatment 6-Pyrotinib
Drug: Dabrafenib+Trametinib — Dabrafenib 150 mg orally twice daily, 28 days as one cycle. Trametinib 150 mg orally twice daily, 28 days as one cycle.
  Arms: Treatment 7-Dabrafenib+Trametinib
Drug: Glecirasib — 800 mg daily orally, 28 days as one cycle.
  Other Names: JAB-21822
  Arms: Treatment 8-Glecirasib
Drug: Ensartinib — 225 mg daily orally, 28 days as one cycle.
  Other Names: X-396
  Arms: Treatment 9-Ensartinib

SUMMARY:
This umbrella trial directed by next generation sequencing (NGS) includes patients with treatment-naive unresectable stage III non-small-cell lung cancer (NSCLC). The aim of the umbrella study is to evaluate the efficacy of induction NGS-directed targeted therapies followed by surgery for stage III NSCLC patients whose tumor harbors a rare mutation.

DETAILED DESCRIPTION:
Stage III non-small-cell lung cancer (NSCLC) patients account for about one-third of newly diagnosed NSCLC, with a large population and strong heterogeneity, posing significant challenges for clinical treatment. Concurrent chemoradiotherapy plus immune checkpoint inhibitors is the recommended therapeutic approach for patients with unresectable stage III non-small cell lung cancer (NSCLC), although surgery offers the chance of cure. However, existing evidence suggests that patients with driver mutation positive NSCLC have limited benefits from immunotherapy. There is still controversy over the definition of 'unresectable', and some stage IIIA and specific stage IIIB-N2 patients may also benefit from comprehensive surgical treatment. Emerging data supports the use of targeted therapies in NSCLC patients with a rare mutation. The aim of this umbrella study is to explore the efficacy of induction next generation sequencing (NGS)-directed targeted therapies followed by surgery for unresectable stage III NSCLC patients whose tumor harbors a rare mutation (Without EGFR Sensitizing Mutations).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have treatment-naive unresectable stage III NSCLC according to the AJCC 8th edition staging;
* Squamous or non-squamous NSCLC histology;
* Subjects should have a rare mutation based on NGS, including mutations of EGFR exon20ins, ROS1 fusion, RET fusion, NTRK fusion, MET 14 exon, HER2, BRAF V600E, KRAS G12C, and ALK fusion.
* Subjects should be without EGFR exon 19 deletions or exon 21 L858R activating mutation;
* Male and female, aged 18-75 years;
* Blood and specimens before and after treatment must be provided;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
* Adequate hematological function: Absolute neutrophil count (ANC) ≥2.0 x 109/L, and Platelet count ≥100 x 109/L, and Hemoglobin ≥9 g/dL (may be transfused to maintain or exceed this level);
* Adequate liver function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN), Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 x ULN;
* Adequate renal function: Serum creatinine ≤ 1.25 x ULN, or ≥ 60 ml/min;
* Female subjects should not be pregnant or breast-feeding;
* Written informed consent provided. Being willing and able to comply with the visits, treatment plan, laboratory examinations and other study procedures scheduled in the study.

Exclusion Criteria:

* Not unresectable stage III disease according to the investigator;
* Subjects with known EGFR sensitive mutations;
* Previous treatment with systemic antitumor therapy for NSCLC;
* Eye inflammation or eye infection not fully treated or conditions predisposing the subject to this.
* History of another malignancy in the last 5 years with the exception of the following: other malignancies cured by surgery alone and having a continuous disease-free interval of 5 years are permitted. Cured basal cell carcinoma of the skin and cured in situ carcinoma of the uterine cervix are permitted.
* Evidence of clinically active interstitial lung disease;
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS);
* Inability to comply with protocol or study procedures;
* Any unstable systemic disease (including active infection, active tuberculosis uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease);
* A serious concomitant systemic disorder that, in the opinion of the investigator, would compromise the patient's ability to complete the study and may confuse the study results;
* Women who are pregnant or nursing.
* Ingredients mixed with small cell lung cancer patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Resectability rate | Baseline to 6 months

SECONDARY OUTCOMES:
Adverse Events | Baseline to 24 months
  Adverse Events were monitored according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0.
Two-year disease-free survival | 2 years after the last patient is randomized
  Disease-free survival was assessed from randomization to disease recurrence or death as a result of any cause.
Two-year overall survival | 2 years after the last patient is randomized
  Overall survival was assessed from randomization to death as a result of any cause.
Number of participants with perioperative complications | Baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Si-Yu Wang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided